CLINICAL TRIAL: NCT04973072
Title: The Effect of Small Wins on Body Fat Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noah Lim (Other)
Responsible Party: Sponsor-Investigator, Noah Lim, Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NUS-IRB-2021-48
Record Dates: First submitted 2021-07-08; First posted 2021-07-22 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants in this arm will not receive any intervention.
- One large reward (Experimental): Participants in this arm will receive S$300 if they reach the PBF goal at the end of 12 weeks.
  Interventions: Behavioral: One large reward treatment
- Small wins (Experimental): Participants in this arm will receive cash rewards capped by S$300, depending on which intermediate goals they reach and the PBF at the end of the 12 weeks.
  Interventions: Behavioral: Small wins treatment

INTERVENTIONS:
Behavioral: One large reward treatment — Participants will be awarded S$300 for reaching the PBF goal at the end of 12 weeks.
  Arms: One large reward
Behavioral: Small wins treatment — The cash rewards that participants will receive are capped by $300 and depend on which IGs they achieve and whether they maintain their progress at the end of the 12 weeks. Specifically, given the PBF goal, the Loss Target (LT) is the difference between the initial PBF measured at the first visit and the PBF goal, i.e., LT = initial PBF - PBF goal. Then, the IG1 is to achieve 25% of the LT, the IG2 is to achieve 50% of the LT, and the IG3 is to achieve 75% of the LT. Participants will earn $75 credits to their accounts on the programme website for reaching each intermediate goal. Also, when they miss IG1 and/or IG3, they can earn the previous missing $75 credits if they reach the IG2 and the LT. At the end of the 12 weeks, they will lose some or all the credits that they have accumulated if they fail to maintain the progress, and they will only receive the corresponding amount in cash
  Arms: Small wins

SUMMARY:
This 24-week-long study compares the effectiveness of two finance incentive structures for weight loss: 1) smaller rewards for achieving intermediate goals vs 2) large reward for achieving an overall goal. Target participants are male Singaporeans or Permanent Residents who are overweight and otherwise healthy.

DETAILED DESCRIPTION:
This study, which spans 24 weeks (12 treatment, 12 post-treatment), aims to compare the effectiveness of 2 financial incentive structures: smaller rewards for achieving intermediate goals vs. a large reward for achieving an overall goal - on weight loss. Male Singaporeans or Permanent Residents between the ages of 25 and 60 will be recruited. Participants must be healthy and have a body mass index (BMI) of between 23 and 27.5, and own and use a smartphone or tablet. Participants will be given an individual-tailored percentage body fat (PBF) goal and will be blinded from the presence of different treatment conditions and randomly assigned to one of the three conditions for 12 weeks:

1. Control group. Participants will receive only participation fees.
2. One large reward treatment. Participants will be awarded S$X for reaching the PBF goal at the end of 12 weeks.
3. Small wins treatment. Participants in the Small wins treatment condition will also be given 3 triweekly intermediate goals (IGs). Specifically, given the PBF goal, the PBF Loss Target (LT) is the difference between the initial PBF measured at the first visit and the goal, i.e., LT = initial PBF - PBF goal. Then, the IG1 is to achieve 25% of the LT, the IG2 is to achieve 50% of the LT, and the IG3 is to achieve 75% of the LT. The cash rewards that participants will receive are capped by S$X and depend on which IGs participants achieve and whether participants maintain their progress at the end of the 12 weeks.

All participants will be given an individual-tailored 12-week percentage body fat (PBF) goal. The formula for this goal will be set in consultation with medical and fitness professionals (including certified doctors and fitness trainers) to ensure that it is safe, challenging, and achievable. The base formula, which assumes a 5% weight loss as is often defined to be the medically significant level, is:

(P* W - x*5%*W)/(95%*W)

where P is PBF at baseline (week 1), W is body mass in kg at baseline, P*W is their body fat mass at baseline, and x, ranging between 0% and 100%, is the parameter that is set in consultation with professionals. At 100%, it implies that all 5% in weight loss is from fat, vice versa.

Because P and W differ between most persons, the formula tailors a different goal to each research subject. The formula is meant to be flexible toward each individual participant's baseline weight and body fat percent. Leveraging the 5% weight loss target, the investigators determined the expected percentage of this weight that is lost as fat, knowing that weight loss includes not only fat loss but also other components such as water loss. In previous studies, for 1 kg loss in weight, on average, 78.8% came from body fat. Hence, the investigators have targeted 80% of weight loss from the participants to come from body fat.

To examine changes in health, objective measurements will be made during scheduled participant visits on Weeks 1, 12, and 24. Measures include height, weight, waist circumference, and PBF. Each participant will also be given a free digital scale for personal use from home. Their weight and PBF data from the scale will be synchronized to a mobile application. The investigators will retrieve with the participant's consent to examine changes throughout the study's duration.

There are a total of 3 scheduled visits. The first in Week 1 allows baseline measures to be determined. During the first visit, the participants will be provided with a Weight Loss Brochure to warn against the harmful effects of excessive weight loss. The second visit in Week 12 marks the end of the treatment and allows treatment effects to be investigated. The last visit in Week 24 checks for post-treatment effects. During all 3 visits, the participants will also complete a Health Risk Assessment Survey. This survey should take no longer than 10 minutes to complete, and the research team will be physically present to assist the participants with it if so required.

Due to the uncertainty of the pandemic, the investigators may hold the second and/or the third research visits virtually (or at least provide an online option) to avoid large gatherings if necessary. For each virtual research visit, the research team will contact the participants through a video call, during which participants will step on the weighing scales and show the readings to the team. If a research visit is held online, the participation fee/rewards will be sent electronically. The research team will still hold physical meetings for those who experience technical difficulties.

To let the participants track their PBF progress, every participant would be given a digital scale for their keeping even after the research has concluded. Referring to the Health Products Act (HPA), this scale would not be defined as a "medical device." The digital scale serves simply, as would a conventional scale, to inform the user on some bodily metric. It does not attempt to make any medical judgment or recommendation for the user. The research team has done testing on the digital scale and is satisfied with the precision of the device. The participants are expected to weigh-in on the scales weekly from home at their convenience. In the middle of each of the 12 weeks (e.g., Wednesday or Thursday), an automated email will be sent to the participants reminding the participants to do so by the end of the week (Sunday). Non-compliance will not be penalized, but participants are strongly encouraged to weigh-in. The following is the complete list of data that the participants will access from the scale's mobile application. The researchers, with the participants' consent, will also retrieve this data for analysis: 1. Basal metabolism rate; 2. BMI; 3. Bone mass; 4. Metabolic age; 5. Muscle mass; 6. PBF; 7. Skeletal muscle weight ratio; 8. Subcutaneous fat; 9. Total body water; 10. Visceral fat; 11. Weight

ELIGIBILITY:
Inclusion Criteria:

* Singaporeans or PRs
* Male
* Between the ages of 25 and 60
* Body mass index (BMI) of between 23 and 27.5
* Own and use a smartphone or tablet

Exclusion Criteria:

* Currently participating in any other research program focused on physical activity or weight loss. Note: exercise or education programs (e.g. gym membership, diabetes education class) do not count as research programs.
* Have any reasons why they would not be able to complete a 24-week research program focused on improving health (e.g., plan to move to another country)
* Have a serious medical condition, including one or more of the following conditions: High blood pressure (hypertension), High cholesterol (Hyperlipidaemia), Heart attack (Myocardial infarction), Heart failure, Stroke (Cerebrovascular disease), Chronic obstructive pulmonary disease (COPD), Kidney disease, and Diabetes (Type 2).

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Whether reaching the prescribed PBF goal | At the end of the 12 weeks
  This is a binary variable, which is 1 if the participant reaches the prescribed PBF goal, and 0 otherwise
Whether maintaining what has achieved in the post-treatment period | At the end of the 24 weeks
  This is a binary variable, which is 1 if the participant loses more fat in the post-treatment period than in the intervention period, and 0 otherwise
Achievement Percentage | At the end of the 12 weeks
  A percentage of the change in PBF from the predetermined change in PBF
Weekly Achievement Percentage | Through the study completion (24 weeks)
  A percentage of the change in PBF from the predetermined change in PBF

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lim, PhD, Study Director — The Global Asia Institute, The National University of Singapore; Alessandro Del Ponte, PhD, Principal Investigator — Institution for Social and Policy Studies, Yale University; Ta-Cheng Huang, PhD, Principal Investigator — The Global Asia Institute, The National University of Singapore; Aidas Masiliunas, PhD, Principal Investigator — The Global Asia Institute, The National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaston TB, Dixon JB, O'Brien PE. Changes in fat-free mass during significant weight loss: a systematic review. Int J Obes (Lond). 2007 May;31(5):743-50. doi: 10.1038/sj.ijo.0803483. Epub 2006 Oct 31. PMID 17075583